CLINICAL TRIAL: NCT07153705
Title: OCS Products Based on Exosome Technology Were Applied in the Recurrence Monitoring Study After the Initial Treatment of Baseline CA125-negative Ovarian Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Beihua Kong (Other)
Responsible Party: Sponsor-Investigator, Beihua Kong, archiater, Shandong University
Organization: Shandong University (Other)
Other Study IDs: CM-2401
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
To study the performance of OCS products based on exosome detection technology in monitoring the recurrence of baseline CA125-negative ovarian cancer patients after initial treatment, and to explore reliable methods for monitoring the recurrence of baseline CA125-negative ovarian cancer patients after initial treatment.

ELIGIBILITY:
Inclusion criteria:

1. Women over 18 years old;
2. Pathologically confirmed as stage I-IV primary epithelial ovarian malignant tumor;
3. ECOG < 2;
4. The expected survival period exceeds 6 months;
5. CA125 ≤ 35 U/ml before initial treatment;
6. Undergo surgery and adjuvant chemotherapy;
7. The period between diagnosis and enrollment does not exceed 8 weeks;
8. Be willing to provide blood samples for OCS testing during the research process;
9. Sign the informed consent form.

Exclusion criteria

1. Have had other malignant tumors within the last five years;
2. Have received any treatment for ovarian cancer;
3. Benign ovarian mass;
4. Non-primary ovarian tumors;
5. Combined with other malignant tumors;
6. Patients receiving neoadjuvant therapy;
7. Pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
OCS product inspection | Before the operation